CLINICAL TRIAL: NCT06459596
Title: Communal Coping Intervention for Adults With Type 2 Diabetes
Brief Title: Pilot Brief Communal Coping Intervention for Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Vicki Helgeson, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY2024_00000148
Record Dates: First submitted 2024-05-07; First posted 2024-06-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communal Coping Intervention (Experimental): Experimental: Communal Coping Intervention
  The intervention consists of a single session brief communal coping intervention followed by 7 days of intervention prompts delivered via text message to help couples generalize what they have learned into their daily life. There are 9 components to the intervention:
  establishment of rapport, shared stressor recollection, communal coping education, application of appraisal to diabetes, we-statements to reframe diabetes as shared, facilitated discussion between couple members to identify each person's needs with active listening, collaborative implementation intentions, EMI (ecological momentary intervention) text messaging for 7 days following intervention
  Interventions: Behavioral: Communal Coping Intervention
- Diabetes Education Attention Control (No Intervention): These participants will receive diabetes education via a 15-20 minute videotape (as well the intervention group)

INTERVENTIONS:
Behavioral: Communal Coping Intervention — The components of the intervention were described in the experimental arm.
  Arms: Communal Coping Intervention

SUMMARY:
The investigators plan to develop a communal coping intervention aimed at instilling a shared appraisal of diabetes and increasing patient-partner collaboration. To that end, the investigators will pilot the first randomized clinical trial of a brief communal coping intervention among couples in which one person has T12

DETAILED DESCRIPTION:
The investigators will recruit 66 couples in which one person has type 2 diabetes. Power is based on effect sizes from previous couple intervention studies and meta-analyses on primary outcomes. Couples will be randomly assigned to either a communal coping intervention or an attention (diabetes education) control group. All couples will come to the laboratory or meet via zoom, complete a baseline questionnaire assessment (primary and secondary outcomes, mediators) and have a videotaped conversation about how they cope with diabetes. The intervention group will receive the communal coping intervention. Couples in the intervention group will identify 5 collaborative implementation intentions, whereas controls will identify 5 individual implementation intentions. After the in-person session, couples will individually complete a daily diary at the end of the day for 14 consecutive days which focuses on daily communication, mood, and patient self-care. During the first 7 days, the intervention group will receive two text messages per day (morning focus on shared appraisal, evening focus on one of collaborative implementation intentions identified during in-person session). An in-person follow-up interview will take place 6 weeks after the initial session, during which primary outcomes, secondary outcomes, and mediators will be assessed and the videotaped conversation repeated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes for one year

  * married or living with someone for at least one year who is willing to participate in the study as the study partner
  * age 18 and over
  * reliable access to the internet at home

Exclusion Criteria:

* Non-English speakers

  * Patient has a major chronic illness that affects daily life more than diabetes (e.g., currently --undergoing treatment for cancer)
  * Partner does not consent to participate in study
  * Partner has diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
diabetes distress | baseline, 2 weeks, 6 weeks
  change in Type 1 Diabetes Distress Scale (Fisher et al., 2015) from baseline to 6 weeks; higher scores = more distress; range 1-6; also change over ecological momentary assessment period change in Type 1 Diabetes Distress Scale (Fisher et al., 2015) from baseline to 6 weeks; higher scores = more distress; range 1-6; also change over ecological momentary assessment period change in Type 1 Diabetes Distress Scale (Fisher et al., 2015) from baseline to 6 weeks; higher scores = more distress; range 1-6; also change over ecological momentary assessment period
self-management | baseline, 2 weeks, 6 weeks
  change in Summary of Diabetes Self-Care Activities from baseline to 6 weeks; higher score = better self-care; range 1-5; also change over ecological momentary assessment period

SECONDARY OUTCOMES:
depressive symptoms | baseline, 2 weeks, 6 weeks
  change in Center for Epidemiological Depression Scale from baseline to 6 weeks; higher numbers = more depressive symptoms; range = 0 to 30; also change over ecological momentary assessment period
life satisfaction | baseline, 2 weeks, 6 weeks
  change in Diener's life satisfaction scale from baseline to 6 weeks; higher numbers= more life satisfaction; range = 1-7; also change over ecological momentary assessment period
relationship quality | baseline, 2 weeks, 6 weeks
  change in Quality of Marriage Index and intimacy subscale from Personal Assessment of Intimacy in Relationships from baseline to 6 weeks; higher numbers = better; range = 1 to 7; also change over ecological momentary assessment period

OTHER OUTCOMES:
self-reports of communal coping, raters coding of communal coping from videotapes, we-talk from brief interview | baseline, 2 weeks, 6 weeks
  change in communal coping from baseline to 6 weeks; higher = more communal coping; range = 0 to 10; also change over ecological momentary assessment period
emotional, instrumental, informational support, criticism, overprotective behavior | baseline, 2 weeks, 6 weeks
  change in social support and negative social interactions from baseline to 6 weeks; higher numbers = more support or more negative interactions; range = 1-7; also change over ecological momentary assessment period
self-report of diabetes communication, videotaped observations | baseline, 2 weeks, 6 weeks
  change in diabetes communication from baseline to 6 weeks; higher numbers = more communication; range = 0 to 10; also change over ecological momentary assessment period
self-efficacy with diabetes management | baseline, 2 weeks, 6 weeks
  change in self-efficacy subscale from Multidimensional Diabetes Questionnaire from baseline to 6 weeks; higher numbers = greater efficacy; range = 0 to 100%; also change over ecological momentary assessment period

CONTACTS AND LOCATIONS:
Overall Officials: Vicki S Helgeson, Ph.D., Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No